CLINICAL TRIAL: NCT04472377
Title: Evaluate the Agreement of High-risk Human Papillomavirus Type Between Self-collected Vaginal Discharge Sample Using "HygeiaTouch Self Sampling Kit for Woman" and Physician Collected Sample From the Cervix
Brief Title: HPV Typing Between Self- and Physician-sampled
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hygeia Touch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HT19-HPV-01
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Human Papillomavirus Infection; Self Sampling; Vaginal Discharge
Keywords: cervical screening; human papillomavirus typing; self sampling
MeSH Terms: conditions — Papillomavirus Infections; Vaginal Discharge

STUDY DESIGN:
Intervention Model Description: Two samples were collected, one by the study investigator using a cervical swab and another one by the patient using the study device immediately after viewing the instruction video and illustration. The association of the self-collected sample and the physician-collected sample was blinded to the laboratory personnel.
Masking Description: the specimen was marked by code which was intended to mask the sample pairing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study population (Experimental): We enroll a total of 1,200 women, as follows,
  1. 120 cases with no history or current cervical intraepithelial lesion or malignancy.
  2. 180 cases with a history of abnormal Pap test including ASCUS, CIN1, or atypical glandular cell.
  3. 240 cases with a history of atypical squamous cells favor HSIL, dysplasia cannot exclude HSIL, CIN2, CIN3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.
  4. 240 cases with current ASCUS, CIN1, or atypical glandular cell.
  5. 420 cases with current abnormal Pap test as atypical squamous cells favor HSIL, dysplasia cannot exclude HSIL, CIN2, CIN3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.
  Interventions: Device: Self sampling kit for collecting discharge from vaginal fornix

INTERVENTIONS:
Device: Self sampling kit for collecting discharge from vaginal fornix — A device to collect exfoliative cells from vaginal fornix that can self-operated with ease and comfort.
  Other Names: Hygeia Touch Self Sampling Kit for Women

SUMMARY:
Hygeia Touch Inc. developed a safe and comfortable vaginal self-sampling device "Hygeia Touch Self Sampling Kit for Women" to self-collect the vaginal discharge sample for high-risk Human Papillomavirus (hrHPV) detection.

This clinical trial aimed to evaluate the agreement of hrHPV detections between vaginal self-sampling using "Hygeia Touch Self Sampling Kit for Women" and physician sampling, and these results will be applied for TFDA registration approval.

DETAILED DESCRIPTION:
Primary end-point:

1. Agreement of hr-HPV types, including types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68, between the physician-collected sample and self-collected sample
2. Agreement of the presence of hr-HPV between the physician-collected sample and self-collected sample

Secondary end-point:

1. Percentage of the valid sample between self-collected and physician-collected specimens
2. Agreement of all (N = 27) HPV types between the paired samples
3. Adverse events associated with sample collection
4. Questionnaire of the appreciation and satisfaction of using self-collecting vaginal discharge sample using "Hygeia Touch Self Sampling Kit for Women" through a short movie and a brief illustration
5. Correlation between histological diagnosis and HPV types

ELIGIBILITY:
Inclusion Criteria:

1. Woman with a uterine cervix, i.e., with no previous total hysterectomy or radiotherapy for cervical tumor. The woman who received subtotal hysterectomy is allowed.

2. Signed informed consent. 3. Fit any one of the following conditions,

1. with no history or current cervical intraepithelial lesion or malignancy.
2. with a history of abnormal Pap test including atypical squamous cells of undetermined significance, cervical intraepithelial neoplasia grade 1, or atypical glandular cell.
3. with a history of atypical squamous cells favor high-grade squamous intraepithelial lesion, dysplasia cannot exclude high-grade squamous intraepithelial lesion, cervical intraepithelial neoplasia grade 2, cervical intraepithelial neoplasia grade 3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.
4. with current atypical squamous cells of undetermined significance, cervical intraepithelial neoplasia grade 1, or atypical glandular cell.
5. with current abnormal Pap test as atypical squamous cells favor high-grade squamous intraepithelial lesion, dysplasia cannot exclude high-grade squamous intraepithelial lesion, cervical intraepithelial neoplasia grade 2, cervical intraepithelial neoplasia grade 3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.

Exclusion Criteria:

1. History of total hysterectomy
2. Pregnant
3. Current cervicitis that requires therapy
4. Received treatment for cervical lesion within 90 days
5. Had undergone radiotherapy or is receiving radiation over the uterus, cervix or vagina
6. Had sexual activity without a condom in 48 hours
7. Excessive vaginal discharge, either in the ovulation period or due to inflammation
8. is undergoing local therapy with an intravaginal tablet or residual drug in the vaginal canal
9. during mense

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Detection of HPV in female genital tract.
Enrollment: 1210 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Hsueh Chou, MBBS, VS, Study Chair — Chang Gung Memorial Hospital
Locations (3):
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
For clinical trial participation.
Supporting Information: SAP, ICF, CSR
Time Frame: 3 months after accepting for report publication
Access Criteria: to the public

REFERENCES:
- [Result] Chou HH, Yang CY, Chao A, Lin H, Lu CH, Ou YC, Hsu ST, Shih YH, Huang HJ, Lin CT, Chen MY, Sun L, Tsai CC, Fu HC, Huang KG, Wu KY, Wu CH, Hsieh WC, Huang YT, Chen LH, Yang LY, Chang WY, Chang TC, Lai CH. Consistency in human papillomavirus type detection between self-collected vaginal specimens and physician-sampled cervical specimens. J Med Virol. 2024 Mar;96(3):e29426. doi: 10.1002/jmv.29426. PMID 38420851
- [Result] Yang CY, Chang TC, Chou HH, Chao A, Hsu ST, Shih YH, Huang HJ, Lin CT, Chen MY, Sun L, Huang KG, Wu KY, Hsieh WC, Huang YT, Chen LH, Lu CH, Lin H, Cheng CM. Evaluation of a novel vaginal cells self-sampling device for human papillomavirus testing in cervical cancer screening: A clinical trial assessing reliability and acceptability. Bioeng Transl Med. 2024 Mar 13;9(4):e10653. doi: 10.1002/btm2.10653. eCollection 2024 Jul. PMID 39036090

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: We enroll a total of 1,200 women, as follows,
  1. 120 cases with no history or current cervical intraepithelial lesion or malignancy.
  2. 180 cases with a history of abnormal Pap test including ASCUS, CIN1, or atypical glandular cell.
  3. 240 cases with a history of atypical squamous cells favor HSIL, dysplasia cannot exclude HSIL, CIN2, CIN3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.
  4. 240 cases with current ASCUS, CIN1, or atypical glandular cell.
  5. 420 cases with current abnormal Pap test as atypical squamous cells favor HSIL, dysplasia cannot exclude HSIL, CIN2, CIN3, cervical carcinoma in situ, squamous cell carcinoma, atypical glandular cells favor neoplasm, adenocarcinoma in situ, or cervical adenocarcinoma.
  Self sampling kit for collecting discharge from vaginal fornix: A device to collect exfoliative cells from vaginal fornix that can self-operated with ease and comfort.
Period: Overall Study
Arm/Group | Study Population
Started | 1210
Completed | 1210
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 1210
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1210
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Agreement in the Detection of High-risk HPV Type in Physician-sampled Specimen and Self-collected Specimen.
Description: Rate of the "agreement". The "agreement" is defined as either (1) presence of any high-risk HPV type in physician collected specimen, and the patient sampled specimen, or (2) absence of high-risk HPV in physician collected specimen and the patient sampled specimen.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Self-collected Specimens: The high-risk HPV test results of the samples collected by the participants
- Physician-sampled Specimens: The high-risk HPV test results of the samples collected by the physician
Arm/Group | Self-collected Specimens | Physician-sampled Specimens
Number analyzed (Participants) | 1170 | 1170
Participants
  Positive | 581 | 611
  Negative | 589 | 559

2. Secondary Outcome: Agreement in HPV Detection Between Physician Collected Sample and Self-collected Sample
Description: Rate of the "agreement". The "agreement" is defined as either (1) presence of any HPV type in physician collected specimen, and the patient sampled specimen, or (2) absence of any HPV in physician collected specimen and the patient sampled specimen.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Self-collected Specimens: The HPV test results of the samples collected by the participants
- Physician-sampled Specimens: The HPV test results of the samples collected by the physician
Arm/Group | Self-collected Specimens | Physician-sampled Specimens
Number analyzed (Participants) | 1170 | 1170
Participants
  Positive | 718 | 720
  Negative | 452 | 450

3. Secondary Outcome: Percentage of a Valid Specimen, According to the Presence of the Beta-globin Gene in Specimens
Description: Percentage of the presence of the beta-globin gene. The ratio could be calculated between self-collected and physician-collected specimens.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Self-collected Specimens: The beta-globin test results of the samples collected by the participants
- Physician-sampled Specimens: The beta-globin test results of the samples collected by the physician
Arm/Group | Self-collected Specimens | Physician-sampled Specimens
Number analyzed (Participants) | 1170 | 1170
Participants | 1170 | 1170

4. Secondary Outcome: Adverse Event From Self Sampling
Description: The number of participants with any adverse event.
Time Frame: within one month after sample collection
Measure: Count of Participants; unit: Participants
Groups:
- Women Participated in Self-sampling: Adverse event reported by women participated in self-sampling
Arm/Group | Women Participated in Self-sampling
Number analyzed (Participants) | 1210
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 months
Groups:
- Participants With Adverse Events: study device-related adverse events
Arm/Group | Participants With Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/1210
Serious Adverse Events (participants affected / at risk) | 0/1210
Other Adverse Events (participants affected / at risk) | 9/1210
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Adverse Events (N=1210)
Perineal pain (Product Issues) | 7
anxiety (Product Issues) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT04472377/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04472377/SAP_001.pdf